CLINICAL TRIAL: NCT02226120
Title: A Multicenter Study to Evaluate Safety and Tolerability in Patients With Chronic Heart Failure and Reduced Ejection Fraction From PARADIGM-HF Receiving Open Label LCZ696
Brief Title: Safety and Tolerability During Open-label Treatment With LCZ696 in Patients With CHF and Reduced Ejection Fraction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLCZ696B2317; 2014-001971-30 (EudraCT Number)
Record Dates: First submitted 2014-08-25; First posted 2014-08-27 (Estimated); Results first posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Chronic Heart Failure With Reduced Ejection Fraction
Keywords: LCZ696; chronic heart failure; ARNI; Congestive heart failure (CHF); heart failure (HF); acute heart failure syndrome; congestive cardiac failure (CCF)
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LCZ696 (Experimental): Angiotensin receptor antagonist neprilysin inhibitor (ARNI) with target dose of 200 mg bid
  Interventions: Drug: LCZ696

INTERVENTIONS:
Drug: LCZ696 — Angiotensin receptor antagonist neprilysin inhibitor (ARNI) with target dose of 200 mg bid

SUMMARY:
The purpose of this study was to collect safety and tolerability data on LCZ696 in eligible PARADIGM-HF patients who received open-label investigational drug. The parent PARADIGM-HF (NCT01035255) trial was terminated early due to compelling efficacy of LCZ696 in patients with heart failure with reduced ejection fraction (HFrEF) after the final pre-specified interim analysis in March 2014.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent for the extension must be obtained before any assessment is performed.
2. Patients who have completed PARADIGM-HF (protocol CLCZ696B2314) and are able to be safely enrolled into the open-label trial as judged by the investigator.

Exclusion Criteria:

1. Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer
2. History of hypersensitivity or allergy to any of the study drugs, drugs of similar chemical classes, ACEIs, ARBs, or NEP inhibitors as well as known or suspected contraindications to LCZ696
3. Known history of angioedema
4. Requirement of simultaneous treatment with both ACEIs and ARBs
5. Current acute decompensated HF (exacerbation of chronic HF manifested by signs and symptoms that may require intravenous therapy)
6. Symptomatic hypotension and/or a SBP < 100 mmHg at Visit 1 (screening)
7. Estimated GFR < 30 mL/min/1.73m^2 as measured by the simplified MDRD formula at Visit 1 (screening)
8. Presence of bilateral renal artery stenosis
9. Serum potassium > 5.2 mmol/L at Visit 1 (screening)
10. Evidence of hepatic disease as determined by any one of the following: AST or ALT values exceeding 3 x ULN at Visit 1, history of hepatic encephalopathy, history of esophageal varices, or history of portacaval shunt
11. Pregnant or nursing (lactating) women
12. Women of child-bearing potential
13. Any condition, not identified in the protocol, that in the opinion of the investigator is likely to prevent the patient from safely tolerating LCZ696 or complying with the requirements of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1980 (Actual)
Dates: Start 2014-10-16 (Actual); Primary Completion 2017-12-28 (Actual); Study Completion 2017-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (321):
- United States (23):
  - Novartis Investigative Site, Huntsville, Alabama
  - Novartis Investigative Site, Muscle Shoals, Alabama
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Oceanside, California
  - Novartis Investigative Site, Palm Springs, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Santa Rosa, California
  - Novartis Investigative Site, Boynton Beach, Florida
  - Novartis Investigative Site, Des Moines, Iowa
  - Novartis Investigative Site, Covington, Louisiana
  - Novartis Investigative Site, Columbia, Maryland
  - Novartis Investigative Site, Saginaw, Michigan
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Fremont, Nebraska
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Rosedale, New York
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Marion, Ohio
  - Novartis Investigative Site, Rapid City, South Dakota
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Livingston, Texas
  - Novartis Investigative Site, Spokane, Washington
  - Novartis Investigative Site, Waukesha, Wisconsin
- Argentina (15):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Ciudad Autonoma de Bs As, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, Quilmes, Buenos Aires
  - Novartis Investigative Site, CABA, Buenos Aires F.D.
  - Novartis Investigative Site, San Salvador de Jujuy, Jujuy Province
  - Novartis Investigative Site, Salta, Salta Province
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Corrientes
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Formosa
  - Novartis Investigative Site, Mendoza
  - Novartis Investigative Site, San Luis
  - Novartis Investigative Site, Santa Fe
  - Novartis Investigative Site, Santiago del Estero
- Belgium (5):
  - Novartis Investigative Site, Brasschaat
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, La Louvière
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Ronse
- Brazil (16):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Brasília, Federal District
  - Novartis Investigative Site, Goiânia, Goiás
  - Novartis Investigative Site, São Luís, Maranhão
  - Novartis Investigative Site, Uberlândia, Mg-cep
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Belém, Pará
  - Novartis Investigative Site, Recife, Pernambuco
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Marília, São Paulo
  - Novartis Investigative Site, Ribeirão Preto, São Paulo
  - Novartis Investigative Site, Santo André, São Paulo
  - Novartis Investigative Site, São José do Rio Preto, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Votuporanga, São Paulo
- Bulgaria (6):
  - Novartis Investigative Site, Haskovo
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Shumen
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
- Canada (8):
  - Novartis Investigative Site, Victoria, British Columbia
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Kitchener, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Weston, Ontario
  - Novartis Investigative Site, Lévis, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, St-Georges Beauce, Quebec
- Novartis Investigative Site, Temuco, Región de la Araucanía, Chile
- Czechia (10):
  - Novartis Investigative Site, Beroun, Czech Republic
  - Novartis Investigative Site, Brandýs nad Labem, Czech Republic
  - Novartis Investigative Site, Liberec V Kristianova, Czech Republic
  - Novartis Investigative Site, Olomouc, Czech Republic
  - Novartis Investigative Site, Prague 10, Vrsovice, Czech Republic
  - Novartis Investigative Site, Třebíč, Czech Republic
  - Novartis Investigative Site, Bílovec, CZE
  - Novartis Investigative Site, Kolín
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Uherské Hradiště
- Denmark (7):
  - Novartis Investigative Site, Copenhagen
  - Novartis Investigative Site, Esbjerg
  - Novartis Investigative Site, Hellerup
  - Novartis Investigative Site, Randers
  - Novartis Investigative Site, Svendborg
  - Novartis Investigative Site, Vejle
  - Novartis Investigative Site, Viborg
- Estonia (2):
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- Novartis Investigative Site, Tampere, Finland
- France (2):
  - Novartis Investigative Site, Montpellier, Herault
  - Novartis Investigative Site, Paris
- Germany (23):
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Bad Homburg
  - Novartis Investigative Site, Bad Krozingen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Buch
  - Novartis Investigative Site, Dessau
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Elsterwerda
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Huy / OT Anderbeck
  - Novartis Investigative Site, Ingelheim
  - Novartis Investigative Site, Kelkheim
  - Novartis Investigative Site, Köthen
  - Novartis Investigative Site, Künzelsau
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Löhne
  - Novartis Investigative Site, Muehlheim An Der Ruhr
  - Novartis Investigative Site, Mühldorf
  - Novartis Investigative Site, Offenbach
  - Novartis Investigative Site, Wermsdorf
  - Novartis Investigative Site, Wetzlar-Naunheim
  - Novartis Investigative Site, Weyhe
- Guatemala (2):
  - Novartis Investigative Site, Guatemala City, Ciudad
  - Novartis Investigative Site, Guatemala City
- Hong Kong (2):
  - Novartis Investigative Site, Hong Kong
  - Novartis Investigative Site, Hong Kong SAR
- Hungary (6):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Nyiregyháza
  - Novartis Investigative Site, Szekszárd
  - Novartis Investigative Site, Székesfehérvár
  - Novartis Investigative Site, Zalaegerszeg
- India (14):
  - Novartis Investigative Site, Guntur, Andhra Pradesh
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Anand, Gujarat
  - Novartis Investigative Site, Surat, Gujarat
  - Novartis Investigative Site, Vadodara, Gujarat
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Ludhiana, Punjab
  - Novartis Investigative Site, Bikaner, Rajasthan
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, Indore
- Israel (7):
  - Novartis Investigative Site, Ashkelon
  - Novartis Investigative Site, Hadera
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Rehovot
  - Novartis Investigative Site, Safed
- Italy (17):
  - Novartis Investigative Site, Aosta, AO
  - Novartis Investigative Site, Cortona, AR
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Treviglio, BG
  - Novartis Investigative Site, Cosenza, CS
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Pozzilli, IS
  - Novartis Investigative Site, Lido di Camaiore, LU
  - Novartis Investigative Site, Milazzo, ME
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Pescia, Point
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Ariccia, RM
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Salerno, SA
  - Novartis Investigative Site, Sassari, SS
- Latvia (2):
  - Novartis Investigative Site, Daugavpils
  - Novartis Investigative Site, Ventspils
- Lithuania (3):
  - Novartis Investigative Site, Kaunas
  - Novartis Investigative Site, Kėdainiai
  - Novartis Investigative Site, Vilnius
- Novartis Investigative Site, Kuala Lumpur, Malaysia
- Mexico (3):
  - Novartis Investigative Site, San Juan del Río, Querétaro
  - Novartis Investigative Site, Aguascalientes
  - Novartis Investigative Site, San Luis Potosí City
- Netherlands (15):
  - Novartis Investigative Site, Breda, CK
  - Novartis Investigative Site, 's-Hertogenbosch
  - Novartis Investigative Site, Amersfoort
  - Novartis Investigative Site, Arnhem
  - Novartis Investigative Site, Blaricum
  - Novartis Investigative Site, Delft
  - Novartis Investigative Site, Ede
  - Novartis Investigative Site, Gorinchem
  - Novartis Investigative Site, Hardenberg
  - Novartis Investigative Site, Harderwijk
  - Novartis Investigative Site, Heerenveen
  - Novartis Investigative Site, Hengelo
  - Novartis Investigative Site, Sneek
  - Novartis Investigative Site, Tilburg
  - Novartis Investigative Site, Veldhoven
- Novartis Investigative Site, Panama City, Panama
- Peru (7):
  - Novartis Investigative Site, Bellavista, Lima region
  - Novartis Investigative Site, Jesus Maria, Lima region
  - Novartis Investigative Site, La Molina, Lima region
  - Novartis Investigative Site, San Borja, Lima region
  - Novartis Investigative Site, San Isidro, Lima region
  - Novartis Investigative Site, San Miguel, Lima region
  - Novartis Investigative Site, Arequipa
- Philippines (4):
  - Novartis Investigative Site, Lipa City, Batangas
  - Novartis Investigative Site, Quezon City, Manila
  - Novartis Investigative Site, Pasig
  - Novartis Investigative Site, Quezon City
- Poland (2):
  - Novartis Investigative Site, Gdynia
  - Novartis Investigative Site, Lublin
- Portugal (7):
  - Novartis Investigative Site, Vila Real, Portuigal
  - Novartis Investigative Site, Covilha
  - Novartis Investigative Site, Guimarães
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Portalegre
  - Novartis Investigative Site, Porto
  - Novartis Investigative Site, Setúbal
- Romania (7):
  - Novartis Investigative Site, Bucharest, District 1
  - Novartis Investigative Site, Craiova, Jud. Dolj
  - Novartis Investigative Site, Timișoara, Timiș County
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Craiova
  - Novartis Investigative Site, Deva
  - Novartis Investigative Site, Timișoara
- Russia (19):
  - Novartis Investigative Site, Ivanovo
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, Kirov
  - Novartis Investigative Site, Krasnodar
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, N.Novgorod
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Novosibirsk-117
  - Novartis Investigative Site, Orenburg
  - Novartis Investigative Site, Perm
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, S-Petersburg
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Smolensk
  - Novartis Investigative Site, Tula
  - Novartis Investigative Site, Vladimir
  - Novartis Investigative Site, Yekaterinburg
- Novartis Investigative Site, Singapore, Singapore
- Slovakia (9):
  - Novartis Investigative Site, Brezno, Slovak Republic
  - Novartis Investigative Site, Košice, Slovak Republic
  - Novartis Investigative Site, Levice, Slovak Republic
  - Novartis Investigative Site, Prešov, Slovak Republic
  - Novartis Investigative Site, Svidník, Slovak Republic
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Lučenec
  - Novartis Investigative Site, Martin
- South Africa (12):
  - Novartis Investigative Site, Bloemfontein, Free State
  - Novartis Investigative Site, Soweto, Gauteng
  - Novartis Investigative Site, Durban, KwaZulu-Natal
  - Novartis Investigative Site, Cape Town, Western Cape
  - Novartis Investigative Site, Alberton
  - Novartis Investigative Site, Bloemfontein
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Durban
  - Novartis Investigative Site, Johannesburg
  - Novartis Investigative Site, Kempton Park
  - Novartis Investigative Site, Pretoria
  - Novartis Investigative Site, Worcester
- South Korea (6):
  - Novartis Investigative Site, Wŏnju, Gangwon-do
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul, Seocho-gu
  - Novartis Investigative Site, Daegu
  - Novartis Investigative Site, Seoul
- Spain (12):
  - Novartis Investigative Site, Marbella, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Sant Joan Despí, Catalonia
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Vigo, Galicia
  - Novartis Investigative Site, Alcalá de Henares, Madrid
  - Novartis Investigative Site, Móstoles, Madrid
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
- Sweden (4):
  - Novartis Investigative Site, Stockholm, SE
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Karlshamn
  - Novartis Investigative Site, Motala
- Taiwan (5):
  - Novartis Investigative Site, Changhua
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Yilan
- Thailand (3):
  - Novartis Investigative Site, Taladkwan, Changwat Nonthaburi
  - Novartis Investigative Site, Muang, Thailand
  - Novartis Investigative Site, Khon Kaen, THA
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Kocaeli
  - Novartis Investigative Site, Sivas
- United Kingdom (27):
  - Novartis Investigative Site, Durham, County Durham
  - Novartis Investigative Site, Dorchester, Dorset
  - Novartis Investigative Site, Basingstoke, Hampshire
  - Novartis Investigative Site, Portsmouth, Hampshire
  - Novartis Investigative Site, Inverness, Invernesshire
  - Novartis Investigative Site, Oldham, Lancashire
  - Novartis Investigative Site, Leicester, Leicestershire
  - Novartis Investigative Site, Craigavon, Northern Ireland
  - Novartis Investigative Site, Dundee, Perthshire
  - Novartis Investigative Site, Taunton, Somerset
  - Novartis Investigative Site, Yeovil, Somerset
  - Novartis Investigative Site, Sheffield, South Yorkshire
  - Novartis Investigative Site, Redhill, Surrey
  - Novartis Investigative Site, South Shields, Tyne and Wear
  - Novartis Investigative Site, Sunderland, Tyne and Wear
  - Novartis Investigative Site, Dudley, West Midlands
  - Novartis Investigative Site, Cheshire
  - Novartis Investigative Site, Coventry
  - Novartis Investigative Site, Exeter
  - Novartis Investigative Site, Kent
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Milton Keynes
  - Novartis Investigative Site, Newport
  - Novartis Investigative Site, Norwich
  - Novartis Investigative Site, Poole
  - Novartis Investigative Site, Rotherham
  - Novartis Investigative Site, Worcester

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 417 sites in 41 countries worldwide.
Pre-assignment Details: The total number in the participant flow and baseline characteristics sections reflects the number of participants treated (1980).
Period: Overall Study
Arm/Group | LCZ696
Started (All enrolled patients who received at least one dose of study medication (Safety Analysis Set (SAF))) | 1980
Completed (Completed open-label treatment) | 1660
Not Completed | 320
Not completed — Adverse Event | 60
Not completed — Death | 172
Not completed — Study terminated by sponsor | 1
Not completed — Technical problems | 4
Not completed — Lost to Follow-up | 13
Not completed — Physician Decision | 21
Not completed — Withdrawal by parent/guardian | 36
Not completed — Non-compliance with study drug | 10
Not completed — Protocol deviation | 1
Not completed — missing treatment disposition pages | 2

BASELINE CHARACTERISTICS:
Arm/Group | LCZ696
Number analyzed (Participants) | 1980
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (10.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 453
  Male | 1527
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 39
  Asian | 305
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 80
  White | 1450
  More than one race | 0
  Unknown or Not Reported | 106

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (AEs), Serious Adverse Events (SAEs) and Deaths as a Measure of Safety and Tolerability of LCZ696
Description: The primary assessments for safety were the reporting of angioedema, AEs suspected to be related to LCZ696, AEs leading to study drug discontinuation and serious adverse events (SAE) including death. The assessment of safety were based primarily on the frequency of adverse events of special interest, sitting systolic and diastolic blood pressure, heart rate, and serious adverse events suspected by the investigators to be related to LCZ696 for the Safety set. Only descriptive analysis done.
Time Frame: From first dose of study treatment to 30 days after last dose of study treatment, up to 30 months.
Population: Safety Set (SAF), which consisted of all enrolled participants who received at least one dose of open-label study medication, was considered. Only descriptive analysis done.
Measure: Count of Participants; unit: Participants
Arm/Group | LCZ696
Number analyzed (Participants) | 1980
Participants
  AEs by Primary System Organ Class (SOC) | 1289
  SAEs by Primary System Organ Class (SOC) | 555
  Deaths by Primary System Organ Class (SOC) | 186

ADVERSE EVENTS:
Time Frame: From first dose of study treatment to 30 days after last dose of study treatment, approximately 30 months
Arm/Group | LCZ696
All-Cause Mortality (participants affected / at risk) | 186/1980
Serious Adverse Events (participants affected / at risk) | 555/1980
Other Adverse Events (participants affected / at risk) | 352/1980
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 (N=1980)
Anaemia (Blood and lymphatic system disorders) | 1
Normocytic anaemia (Blood and lymphatic system disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 3
Acute left ventricular failure (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 9
Adams-Stokes syndrome (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 14
Angina unstable (Cardiac disorders) | 10
Arrhythmia (Cardiac disorders) | 4
Atrial fibrillation (Cardiac disorders) | 14
Atrioventricular block complete (Cardiac disorders) | 5
Bradycardia (Cardiac disorders) | 3
Cardiac arrest (Cardiac disorders) | 13
Cardiac failure (Cardiac disorders) | 144
Cardiac failure acute (Cardiac disorders) | 21
Cardiac failure chronic (Cardiac disorders) | 32
Cardiac failure congestive (Cardiac disorders) | 20
Cardio-respiratory arrest (Cardiac disorders) | 7
Cardiogenic shock (Cardiac disorders) | 8
Cardiorenal syndrome (Cardiac disorders) | 1
Cardiovascular disorder (Cardiac disorders) | 1
Congestive cardiomyopathy (Cardiac disorders) | 4
Cor pulmonale (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 2
Left ventricular dysfunction (Cardiac disorders) | 2
Left ventricular failure (Cardiac disorders) | 4
Myocardial infarction (Cardiac disorders) | 16
Myocardial ischaemia (Cardiac disorders) | 2
Nodal rhythm (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Sinus node dysfunction (Cardiac disorders) | 2
Supraventricular tachycardia (Cardiac disorders) | 1
Systolic dysfunction (Cardiac disorders) | 1
Ventricular arrhythmia (Cardiac disorders) | 5
Ventricular fibrillation (Cardiac disorders) | 5
Ventricular tachycardia (Cardiac disorders) | 31
Phimosis (Congenital, familial and genetic disorders) | 1
Vertigo (Ear and labyrinth disorders) | 2
Adrenal insufficiency (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Cataract (Eye disorders) | 1
Open angle glaucoma (Eye disorders) | 1
Refraction disorder (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 9
Abdominal pain upper (Gastrointestinal disorders) | 3
Ascites (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Diverticulum intestinal (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Duodenitis (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Ileus paralytic (Gastrointestinal disorders) | 1
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 2
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1
Large intestine polyp (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Pancreatic mass (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 3
Cardiac death (General disorders) | 4
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 1
Death (General disorders) | 3
General physical health deterioration (General disorders) | 1
Malaise (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 7
Non-cardiac chest pain (General disorders) | 4
Oedema peripheral (General disorders) | 3
Sudden cardiac death (General disorders) | 15
Sudden death (General disorders) | 13
Bile duct obstruction (Hepatobiliary disorders) | 1
Cholangitis (Hepatobiliary disorders) | 3
Cholecystitis (Hepatobiliary disorders) | 3
Cholecystitis acute (Hepatobiliary disorders) | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 2
Hepatic congestion (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Abdominal sepsis (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 3
Arthritis bacterial (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Bursitis infective (Infections and infestations) | 1
Campylobacter gastroenteritis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 2
Cholecystitis infective (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Diabetic foot infection (Infections and infestations) | 1
Diarrhoea infectious (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 3
Ecthyma (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 2
Gangrene (Infections and infestations) | 3
Gastroenteritis (Infections and infestations) | 5
Hepatitis E (Infections and infestations) | 1
Hepatitis viral (Infections and infestations) | 1
Implant site infection (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Infectious pleural effusion (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Intervertebral discitis (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 4
Lung infection (Infections and infestations) | 1
Orchitis (Infections and infestations) | 2
Otitis media chronic (Infections and infestations) | 1
Ovarian abscess (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 4
Pneumococcal sepsis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 47
Postoperative wound infection (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 3
Sepsis (Infections and infestations) | 12
Sepsis syndrome (Infections and infestations) | 1
Septic shock (Infections and infestations) | 10
Stoma site infection (Infections and infestations) | 1
Streptococcal bacteraemia (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Tracheobronchitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 10
Urosepsis (Infections and infestations) | 3
Viral diarrhoea (Infections and infestations) | 1
Viral infection (Infections and infestations) | 2
Wound sepsis (Infections and infestations) | 1
Chest injury (Injury, poisoning and procedural complications) | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1
Electric shock (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 2
Femur fracture (Injury, poisoning and procedural complications) | 5
Fibula fracture (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Fractured skull depressed (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 3
Humerus fracture (Injury, poisoning and procedural complications) | 1
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 3
Road traffic accident (Injury, poisoning and procedural complications) | 2
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 3
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 2
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1
Arteriogram coronary (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Blood potassium decreased (Investigations) | 1
Blood potassium increased (Investigations) | 2
Ejection fraction abnormal (Investigations) | 1
Functional residual capacity decreased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 2
International normalised ratio increased (Investigations) | 1
Liver function test increased (Investigations) | 1
Weight decreased (Investigations) | 2
Dehydration (Metabolism and nutrition disorders) | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 4
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2
Diabetic complication (Metabolism and nutrition disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Aphasia (Nervous system disorders) | 1
Brain injury (Nervous system disorders) | 1
Brain oedema (Nervous system disorders) | 1
Cerebellar infarction (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 2
Cerebral infarction (Nervous system disorders) | 6
Cerebral ischaemia (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 13
Cervicogenic vertigo (Nervous system disorders) | 1
Coma (Nervous system disorders) | 1
Dementia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 4
Dysarthria (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Facial paralysis (Nervous system disorders) | 1
Haemorrhagic stroke (Nervous system disorders) | 1
Hemianaesthesia (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1
Ischaemic cerebral infarction (Nervous system disorders) | 2
Ischaemic stroke (Nervous system disorders) | 7
Loss of consciousness (Nervous system disorders) | 2
Post stroke seizure (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 2
Radiculopathy (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 7
Transient ischaemic attack (Nervous system disorders) | 4
Device battery issue (Product Issues) | 3
Device malfunction (Product Issues) | 1
Lead dislodgement (Product Issues) | 1
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Disorientation (Psychiatric disorders) | 1
Mental disorder (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 18
Chronic kidney disease (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Leukocyturia (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 12
Renal impairment (Renal and urinary disorders) | 8
Urethral stenosis (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 2
Acquired hydrocele (Reproductive system and breast disorders) | 1
Acquired phimosis (Reproductive system and breast disorders) | 1
Genital ulceration (Reproductive system and breast disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1
Bronchial oedema (Respiratory, thoracic and mediastinal disorders) | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 8
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 2
Treatment noncompliance (Social circumstances) | 1
Aortic aneurysm (Vascular disorders) | 2
Aortic embolus (Vascular disorders) | 1
Circulatory collapse (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Diabetic vascular disorder (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 18
Leriche syndrome (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 2
Peripheral artery occlusion (Vascular disorders) | 1
Peripheral artery stenosis (Vascular disorders) | 1
Peripheral artery thrombosis (Vascular disorders) | 1
Shock (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 (N=1980)
Hyperkalaemia (Metabolism and nutrition disorders) | 118
Hypotension (Vascular disorders) | 252

LIMITATIONS AND CAVEATS:
Two patients had missing treatment epoch disposition pages but were included in Safety Analysis Set (SAF)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-03-02): https://cdn.clinicaltrials.gov/large-docs/20/NCT02226120/SAP_000.pdf
  • Study Protocol (2015-04-28): https://cdn.clinicaltrials.gov/large-docs/20/NCT02226120/Prot_001.pdf